CLINICAL TRIAL: NCT01595035
Title: A Randomized Clinical Trial of a Psycho-educational Intervention to Improve Pain Management After Day Surgery
Brief Title: A Clinical Trial of a Psycho-educational Intervention to Improve Pain Management After Day Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Collaborators: Oslo University Hospital (Other); Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2011/1984
Record Dates: First submitted 2012-05-07; First posted 2012-05-09 (Estimated); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Postoperative Pain; Chronic Pain
Keywords: Day surgery; Orthopedic surgery; Breast reconstruction surgery
MeSH Terms: conditions — Pain, Postoperative; Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- counselling (Experimental): Patients who receive the Pain booklet and support by telephone
  Interventions: Behavioral: psychoeducational
- Control (No Intervention): Standard care

INTERVENTIONS:
Behavioral: psychoeducational — Patients randomized to the intervention group will receive written information about pain and pain treatment in a booklet before surgery and contacted by telephone 24, 48, 72 hours and 7 days after surgery to be coached in pain management
  Arms: counselling

SUMMARY:
Evidence indicates that postoperative pain after day surgery is inadequately controlled. Patients have different experiences and knowledge about how to deal with pain, and the need for information and clarification may vary. The aim of this study is to enhance pain management by academic detailing (patients' current knowledge and motivations are the basis for information) and nurse coaching (frequent and individualized support). The study consists of 4 phases; (1) a pilot study about patients experience with pain after surgery by a structured telephone interview; (2) development of an intervention to improve pain management; (3) implement and evaluate the intervention; (4) evaluate the incidence of chronic pain after day surgery. Even if patients are prescribed sufficient doses of analgesics, pain relief is dependent on patients' adherence with the analgesic regimen. Psychological factors, such as catastrophizing may also contribute to patients' experience of postoperative pain. Strategies that may be more effective than general information concerning surgery and pain management is academic detailing and nurse coaching, and will be used as frame for the intervention.

Hypothesis:

Over the seven days after surgery patients in the intervention group report;

* higher adherence with the analgesic regimen,
* have less pain intensity and pain interference with function and
* lower severity of side effects compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age;
* able, to read, write, and understand Norwegian;
* are scheduled for orthopedic (shoulder, bunnies), or breast reconstruction surgery and
* have a telephone line.

Exclusion Criteria:

* Staying overnight in hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-05; Primary Completion 2020-02 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Average pain intensity | 1 week
  Brief Pain Inventory

SECONDARY OUTCOMES:
The relationships between pain sensitivity, catastrophizing, perceived barriers to pain management and adherence to analgesics and pain intensity. | 1,2,3,7 day after surgery
Pain occurence | 3 and 6 month after surgery
  Brief Pain Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Berit Valeberg, PhD, Principal Investigator — Oslo Metropolitan University
Locations (1):
- Oslo and Akershus University College of Apllied Sciences, Oslo, Norway

REFERENCES:
- [Derived] Valeberg BT, Dihle A, Smastuen MC, Endresen AO, Rustoen T. The effects of a psycho-educational intervention to improve pain management after day surgery: A randomised clinical trial. J Clin Nurs. 2021 Apr;30(7-8):1132-1143. doi: 10.1111/jocn.15659. Epub 2021 Jan 25. PMID 33432643